CLINICAL TRIAL: NCT05020067
Title: Impact on Xerostomia for Nasopharyngeal Carcinoma Patients Treated With or Without Superficial Parotid Lobe-sparing Intensity-modulated Radiotherapy: a Prospective Phase II Clinical Randomized Controlled Study
Brief Title: Impact on Xerostomia for Nasopharyngeal Carcinoma Patients Treated With or Without Superficial Parotid Lobe-sparing Intensity-modulated Radiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPLS-IMRT NPC
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Nasopharyngeal Carcinoma; Radiation-induced Xerostomia
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPLS-IMRT (Experimental): The superficial parotid lobe was contoured as an OAR, and V26 (the percentage volume receiving 26 Gy or more) in the superficial parotid lobe was constrained to be less than 30%
  Interventions: Radiation: superficial parotid lobe-sparing intensity-modulated radiotherapy
- C-IMRT (No Intervention): The entire parotid gland was delineated as an OAR, and V36 (the percentage volume receiving 36 Gy or more) in the entire parotid gland was constrained to be less than 40%

INTERVENTIONS:
Radiation: superficial parotid lobe-sparing intensity-modulated radiotherapy — The superficial parotid lobe was contoured as an OAR, and V26 (the percentage volume receiving 26 Gy or more) in the superficial parotid lobe was constrained to be less than 30%.
  Arms: SPLS-IMRT

SUMMARY:
This is a prospective phase II clinical randomized controlled study, the purpose of this study is to assess whether superficial parotid lobe-sparing intensity-modulated radiotherapy (SPLS-IMRT) can decrease the incidence of xerostomia versus conventional IMRT (C-IMRT) in NPC patients.

ELIGIBILITY:
Inclusion Criteria:1) newly diagnosed, histologically confirmed World Health Organization (WHO) type II-III NPC; 2) stage I-IVa (T1-4 N0-3M0) according to the staging system of the 8th American Joint Committee on Cancer/Union for International Cancer Control (AJCC/UICC); 3) no prior antitumor therapy; 4) no tumor involvement in salivary gland; 5) no parotid glands disorder and no history of parotid glands surgery; 6) ages between 18 and 70 years; 7) Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, and 8) adequate organ function Exclusion Criteria: 1) used salivary stimulating or protecting agent; 2) metachronous or synchronous malignancy; 3) pregnancy or lactation; or 4) severe comorbidities. The pretreatment evaluation included a complete history and physical examination, nasopharyngoscopy, chest X-ray, complete blood count, liver and renal biochemistry, and magnetic resonance imaging (MRI) of the head and neck.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
the incidence of xerostomia | 12 months
  the incidence of xerostomia at 12m post-RT based on Radiation Therapy Oncology Group (RTOG) criteria

SECONDARY OUTCOMES:
xerostomia questionnaire score | 12 months
  The XQ consisted of 8 specific questions which were listed as follows: difficulty in talking; difficulty in chewing; difficulty in swallowing solid food; frequency of sleeping problems; mouth and throat dryness when eating food; mouth and throat dryness while not eating; frequency of sipping liquids to aid swallowing food; frequency of sipping liquids for oral comfort when not eating.
Salivary flow rate | 12 months
  unstimulated salivary flow rateand stimulated salivary flow rate
locoregional relapse-free survival | 36 months
distant metastasis-free survival | 36 months
overall survival | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang H, Miao J, Xiao X, Hu J, Zhang G, Peng Y, Lu S, Liang Y, Huang S, Han F, Deng X, Zhao C, Wang L. Impact on xerostomia for nasopharyngeal carcinoma patients treated with superficial parotid lobe-sparing intensity-modulated radiation therapy (SPLS-IMRT): A prospective phase II randomized controlled study. Radiother Oncol. 2022 Oct;175:1-9. doi: 10.1016/j.radonc.2022.07.006. Epub 2022 Jul 8. PMID 35817320
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn